CLINICAL TRIAL: NCT00285454
Title: A Phase I/II, Randomised, Double-blind, Placebo Controlled, Single-centre Study of Bone Marrow Mononuclear Cells by Percutaneous Retrograde Coronary Venous Delivery to Patients With Ischaemic Heart Failure and no Standard Revascularisation Options.
Brief Title: Cell Repair in Heart Failure
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no funding
Sponsor: Imperial College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Amanda Heinl-Green
Record Dates: First submitted 2006-01-27; First posted 2006-02-02 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Ischemia
MeSH Terms: conditions — Heart Failure; Ischemia

INTERVENTIONS:
Procedure: Retrograde coronary venous delivery of cells.

SUMMARY:
Many people in the UK have ischaemic heart disease. Insufficient blood supply to the heart muscle means that it functions inefficiently, and leads to symptoms of shortness of breath, chest pain and excess fluid in the body. Recently it has been shown that cells from the inside of bone are able to produce many different cell types. We are investigating a new treatment in which a patient's bone marrow cells are taken, and injected into the heart in an attempt to produce new blood vessels and heart muscle cells. This may lead to a new treatment for ischaemic heart disease.

DETAILED DESCRIPTION:
Study Objectives:

1. Evaluate the safety of a single administration of bone marrow mononuclear cells by retrograde coronary venous delivery.
2. Evaluate the bioactivity of bone marrow mononuclear cells in mediating increased perfusion in viable underperfused areas of myocardium.
3. Evaluate the ability of bone marrow mononuclear cells to improve myocardial function specifically regional wall motion and cardiac synchronisation.
4. Evaluate the use of potential bioactivity assays and clinical outcomes for assessing bone marrow mononuclear cell- induced myocardial changes.

Study Design:

A phase I/II, randomised, double-blind, placebo controlled, single-centre study of bone marrow mononuclear cells by percutaneous retrograde coronary venous delivery to patients with ischaemic heart failure and no standard revascularisation options.

Study Population:

Patients with symptomatic ischaemic heart failure, not amenable to conventional revascularisation strategies (PCI, CABG, LVAD) or transplantation.

Independent Eligibility:

The results of the screening procedures will be compiled and submitted to an independent interventional cardiologist and cardiac surgeon who are not associated with the study for consideration for enrolment. It will be the independent reviewer's responsibility to confirm eligibility prior to a patient participating in the study.

Product:

Autologous bone marrow mononuclear, the first 6 safety and feasibility patients (open-labelled) will receive a sub-population of Indium-111 labelled cells to assess feasibility of delivery. The remaining patients will either receive Active: Bone marrow mononuclear cells and 5 % HSA Placebo: 5% HSA

Route:

Retrograde coronary venous delivery The total dose of bone marrow mononuclear cells or placebo will be divided into two, each administered as a 10ml bolus into a selective coronary veins. There will be significant patient heterogeneity regarding size of ischaemic viable territory present and anatomy of venous system. We aim to treat two veins, individual SPECT and venogram results will be used to direct the venous anatomy to be targeted. An attempt will be made to cover as large an area as possible of a patient's ischaemic viable territory. The total dose of cells will remain constant between patients.

Safety:

The first 6 patients will receive cells as an adjunct to Cardiac resynchronization Therapy and ICD. An external Data Safety and Monitoring Board has also been appointed to oversee this study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic ischaemic multi-vessel coronary artery disease (CAD) not suitable for standard revascularization procedures such as CABG, PCI, LVAD, or heart transplant.
2. Area of reversible inducible ischaemia (>10% of LV on SPECT) performed not more than six months prior to study treatment.
3. LVEF < 45% on optimal medical therapy.
4. NYHA class II- IV patient stable on optimal medical therapy for at least 30 days.
5. Written informed consent and agree to attend hospital appointments for 1 year.
6. Male and females 18 to 80 years of age.

Exclusion Criteria:

1. Left ventricular aneurysm or thrombus.
2. Thoracic aortic aneurysm.
3. Congenital Heart disease
4. Acute unstable angina, idiopathic cardiomyopathy, life-threatening ventricular arrhythmias, recent (less than 6 weeks).
5. Contraindication to MRI or any other study procedure.
6. Presence or history of cancer (except low grade and fully resolved non-melanoma skin malignancy).
7. Any co-morbidity likely to reduce short- term survival or which may interfere with functional testing.
8. Recent myocardial infarction < 6mths.
9. Cerebral vascular accident < 6mths.
10. Active hepatitis, receiving immunosuppressive therapy, undergoing haemodialysis.
11. Clinically significant abnormal haematology.
12. Recent history of alcoholism, drug abuse, or severe emotional, behavioural, or psychiatric problems.
13. Fertile women who are pregnant, nursing, or using no form of contraception.
14. Receiving experimental medications or participating in another study within 12 weeks of enrolment into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2006-02 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Safety: up to one year
Efficacy
Co-primary endpoints at 180 Days
Perfusion (MIBI SPECT)
Function (CMR)

SECONDARY OUTCOMES:
Efficacy: at 180 days
Perfusion (CMR)
Function (ECHO, SPECT)
Exercise (VO2 Max)
QOL

CONTACTS AND LOCATIONS:
Overall Officials: Eric WF Alton, Principal Investigator — The Department of Gene Therapy, The NHLI Imperial College London; Jonathan R Clague, Principal Investigator — The Royal Brompton Hospital London
Locations (1):
- The Department of Gene Therapy, The National Heart and Lung Institute, Imperial College London and The Royal Brompton Hospital., London, Middlesex, United Kingdom